CLINICAL TRIAL: NCT01017835
Title: Simvastatin in the Treatment of Isolated Arterial hyPertension and Prevention of cARdiovascular Events
Brief Title: Simvastatin in Patients With Isolated Arterial Hypertension
Acronym: STIPPARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Maciej Banach, Departament of Hypertension
Other Study IDs: 503-5139-2
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension
Keywords: statins; isolated hypertension; atherosclerosis; lipid profile
MeSH Terms: conditions — Hypertension; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- statin treatment, isolated hypertension: treatment with statins, patients with isolated hypertension, with no hyperlipidemia, no diabetes, no smoking
- placebo treatment, isolated hypertension: treatment with placebo, patients with isolated hypertension, with no hyperlipidemia, no diabetes, no smoking

SUMMARY:
The purpose of this study is to determine whether combined therapy with simvastatin and hypotensive drugs (ACEI or ARB) may decrease the blood pressure. Moreover, we would like to assess the influence of isolated hypertension on endothelial injury, and on the development of atherosclerosis.

DETAILED DESCRIPTION:
Hypertension is one of the most important predictors of cardiovascular diseases (CVD). Due to the fact that hypertension frequently coexists with hypercholesterolemia and diabetes which increase the risk of CVDs development, it is advisable to use the optimal combined therapy (hypotensive + hypolipidemic + hypoglycemic)in this group of patients. Statins are the most effective and widely used drugs for the treatment of hypercholesterolemia. According to the available experimental and clinical data they may decrease the blood pressure (BP) in normotensive and hypertensive patients. However, it is still difficult to determine to what degree the reduction of both blood pressure and cardiovascular risk is due to hypotensive or hypolipidemic/pleiotropic effects of statins.

ELIGIBILITY:
Inclusion Criteria:

* isolated hypertension (I or II class according to ESH guidelines 2009)

Exclusion Criteria:

* ischemic heart disease, prior percutaneous coronary intervention (PCI), prior coronary artery bypass grafting (CABG), heart failure, diabetes, hyperlipidemia, active smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the Department of Nephrology, Hypertension and Family Medicine,Clinical Hospital of Medical University of Lodz
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Banach, MD PhD, Study Chair — Departament of Hypertension , Medical University of Lodz
Locations (1):
- Departament of Nephrology, Hypertension and Family Medicine, Clinical Hospital of Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Background] Stepien M, Banach M, Mikhailidis DP, Gluba A, Kjeldsen SE, Rysz J. Role and significance of statins in the treatment of hypertensive patients. Curr Med Res Opin. 2009 Aug;25(8):1995-2005. doi: 10.1185/03007990903098081. PMID 19555312
- [Background] Rysz J, Aronow WS, Stolarek RS, Hannam S, Mikhailidis DP, Banach M. Nephroprotective and clinical potential of statins in dialyzed patients. Expert Opin Ther Targets. 2009 May;13(5):541-50. doi: 10.1517/14728220902882130. PMID 19368496
- [Background] Szadkowska I, Stanczyk A, Aronow WS, Kowalski J, Pawlicki L, Ahmed A, Banach M. Statin therapy in the elderly: a review. Arch Gerontol Geriatr. 2010 Jan-Feb;50(1):114-8. doi: 10.1016/j.archger.2008.12.012. Epub 2009 Feb 13. PMID 19217673